CLINICAL TRIAL: NCT03773445
Title: Association of Golimumab Trough Levels With Endoscopic and Histologic Healing in Patients With Ulcerative Colitis
Brief Title: Golimumab Trough Levels in Patients With Ulcerative Colitis
Acronym: GLMLEVEL
Status: Completed | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Hospital Universitario La Fe (Other); Hospital Universitario 12 de Octubre (Other); Hospital Universitario Ramon y Cajal (Other); Gregorio Marañón Hospital (Other); Complejo Hospitalario de Navarra (Other); Hospital Universitario Fundación Alcorcón (Other); Hospital Infanta Sofia (Other); Hospital Clínico Universitario de Valencia (Other); Puerta de Hierro University Hospital (Other); Hospital Universitario La Paz (Other); Hospital Universitario de Fuenlabrada (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Carlos Taxonera, Dr., Hospital San Carlos, Madrid
Other Study IDs: CTS-GOL-2018-01
Record Dates: First submitted 2018-11-25; First posted 2018-12-12 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; golimumab; simponi; therapeutic drug monitoring; endoscopic healing; histologic remission
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Shadowing Technique, Histology; Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and colonic biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Golimumab trough levels — Golimumab trough levels taken immediately before the administration of the next subcutaneous dose of golimumab
Diagnostic Test: Antibodies to golimumab — Antibodies to golimumab taken immediately before the administration of the next subcutaneous dose of golimumab
Diagnostic Test: Histology — Histology of colonic biopsies using the Geboes Index
Diagnostic Test: Colonoscopy — Colonoscopy to evaluate the endoscopic activity by a Mayo endoscopic subscore

SUMMARY:
Proactive therapeutic drug monitoring of Anti-TNFs with drug titration to a therapeutic window is associated with favorable long-term therapeutic outcomes in IBD and may be superior to reactive therapeutic drug monitoring. Moreover, many exposure-response relationship studies have shown that higher serum anti-TNF drug concentrations are associated with better clinical outcomes in IBD, suggesting that it is maybe time to go from a 'treat-to-target' to a 'treat-to trough' therapeutic approach. In this scenario, there are very limited data regarding therapeutic drug monitoring with golimumab in UC and even no data regarding a therapeutic window to target for important objectives outcomes like mucosal healing and histological remission.

DETAILED DESCRIPTION:
Tumor necrosis factor (TNF)-α antagonists have changed the goals of ulcerative colitis (UC) treatment, with the focus now on preventing disease progression rather than just controlling symptoms. Anti-TNF agents have shown ability to achieve clinical remission and mucosal healing in UC. However, histological remission represents a target distinct from endoscopic healing in UC, and seems a better predictor of clinical outcomes. Moreover, histological remission and not mucosal healing has been associated with a reduced risk of colorectal cancer in UC. Infliximab was reported to induce histological remission in a significant proportion of UC patients. More recently, adalimumab was able to achieve histological remission in nearly one-third of anti-TNF naïve patients with moderately to severely active UC.

Reactive therapeutic drug monitoring of anti-TNF agents may help to identify mechanisms for loss of response and to guide selection of optimal intervention in individual patients and has been shown to be cost-effective compared with empiric dose escalation. Proactive therapeutic drug monitoring showed that anti-TNF trough levels are correlated with clinical response, clinical remission and mucosal healing in patients with inflammatory bowel disease (IBD). Conversely, inadequate serum drug concentrations and antidrug antibodies are associated with poor clinical outcomes. Recently, a study demonstrated that infliximab trough concentrations during maintenance therapy are associated with endoscopic and histologic healing in patients with UC.

Golimumab, a subcutaneously administered fully human antibody to TNF, induces clinical response and remission in patients with moderately to severely active UC. In patients who responded to induction therapy, golimumab doses administered every 4 weeks as a maintenance regimen was effective in maintaining clinical response through 1 year. Available data on golimumab drug monitoring and exposure-response relationship in UC patients are from the PURSUIT trials. A positive association between golimumab levels and efficacy outcomes, including mucosal healing, was confirmed during both induction and maintenance portions of the PURSUIT studies.

Real life data regarding golimumab concentrations and clinical outcomes are lacking, with only a small observational study published. Besides, there are no data regarding the ability of golimumab to achieve histological remission in UC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Patients with a diagnosis of ulcerative colitis at least 12 months prior to the start of the study.
* Patients previously treated with golimumab for ulcerative colitis prescribed according to the usual clinical practice of each center and who have received at least 5 maintenance doses according to the guidelines accepted in the technical file.
* Sign of informed consent.

Exclusion Criteria:

* Patients with Crohn's disease or colitis pending classification
* Alterations in the coagulation that contraindicate the taking of biopsies
* Patients with moderate-severe heart failure (grades III / IV NYHA)
* Patients with tuberculosis or other serious infections such as septicemia, abscesses and opportunistic infections
* Psychiatric illness that discourages participation in the study
* Patients with a history of hypersensitivity to golimumab, to other murine proteins or to any of the excipients included in the golimumab data sheet
* Withdrawal of the informed consent by the patient
* Any other condition that in the opinion of the investigator discourages the participation of the subject in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will include patients of at least 18 years old with moderate to severe UC treated with maintenance therapy with golimumab according to usual clinical practice and have received the induction regimen with the drug according to the EU label, followed by maintenance treatment for at least 6 months from the first dose of drug.
  The study population will comprise all consecutive patients in which a programmed colonoscopy is indicated according to clinical practice for one of the following reasons:
  1. Based on a treat-to-target strategy
  2. Screening for prevention of colorectal cancer ( >8 years disease)
  3. In case of flare
  4. In case of long term remission
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between Golimumab trough levels and Endoscopic remission | Cross-Sectional: 15 days before or after the extraction of levels
  defined as a Mayo endoscopic subscore of 0
Correlation between Golimumab trough levels and Endoscopic healing | Cross-Sectional: 15 days before or after the extraction of levels
  defined as a Mayo endoscopic subscore of 0 or 1
Correlation between Golimumab trough levels and Histological remission | Cross-Sectional: 15 days before or after the extraction of levels
  defined as a Geboes index ≤3.0

SECONDARY OUTCOMES:
Correlation between Golimumab trough levels and Clinical remission | Cross-Sectional: 15 days before or after the extraction of levels
  defined as a total Mayo score ≤2 with no individual subscore exceeding 1 point
Correlation between Golimumab trough levels and Clinical response | Cross-Sectional: 15 days before or after the extraction of levels
  defined as a decrease from baseline in the total Mayo score of at least 3-points
Receiver operating characteristic curve analysis | Cross-Sectional: 15 days before or after the extraction of levels
  Thresholds of golimumab levels for outcomes 1 to 5 will be determined using the receiver operating characteristic curve analysis.
C-reactive protein and fecal calprotectin. | Cross-Sectional: 15 days before or after the extraction of levels
  Correlation between Golimumab trough levels with C-reactive protein and fecal calprotectin.
Histological remission | Cross-Sectional: 15 days before or after the extraction of levels
  Proportion of patients with Histological remission defined as a Geboes index ≤3.0

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Taxonera, Dr., Principal Investigator — Hospital San Carlos, Madrid
Locations (12):
- Spain (12):
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Result] Sandborn WJ, van Assche G, Reinisch W, Colombel JF, D'Haens G, Wolf DC, Kron M, Tighe MB, Lazar A, Thakkar RB. Adalimumab induces and maintains clinical remission in patients with moderate-to-severe ulcerative colitis. Gastroenterology. 2012 Feb;142(2):257-65.e1-3. doi: 10.1053/j.gastro.2011.10.032. Epub 2011 Nov 4. PMID 22062358
- [Result] Sandborn WJ, Feagan BG, Marano C, Zhang H, Strauss R, Johanns J, Adedokun OJ, Guzzo C, Colombel JF, Reinisch W, Gibson PR, Collins J, Jarnerot G, Hibi T, Rutgeerts P; PURSUIT-SC Study Group. Subcutaneous golimumab induces clinical response and remission in patients with moderate-to-severe ulcerative colitis. Gastroenterology. 2014 Jan;146(1):85-95; quiz e14-5. doi: 10.1053/j.gastro.2013.05.048. Epub 2013 Jun 2. PMID 23735746
- [Result] Rosenberg L, Nanda KS, Zenlea T, Gifford A, Lawlor GO, Falchuk KR, Wolf JL, Cheifetz AS, Goldsmith JD, Moss AC. Histologic markers of inflammation in patients with ulcerative colitis in clinical remission. Clin Gastroenterol Hepatol. 2013 Aug;11(8):991-6. doi: 10.1016/j.cgh.2013.02.030. Epub 2013 Apr 13. PMID 23591275
- [Result] Zenlea T, Yee EU, Rosenberg L, Boyle M, Nanda KS, Wolf JL, Falchuk KR, Cheifetz AS, Goldsmith JD, Moss AC. Histology Grade Is Independently Associated With Relapse Risk in Patients With Ulcerative Colitis in Clinical Remission: A Prospective Study. Am J Gastroenterol. 2016 May;111(5):685-90. doi: 10.1038/ajg.2016.50. Epub 2016 Mar 15. PMID 26977756
- [Result] Bryant RV, Burger DC, Delo J, Walsh AJ, Thomas S, von Herbay A, Buchel OC, White L, Brain O, Keshav S, Warren BF, Travis SP. Beyond endoscopic mucosal healing in UC: histological remission better predicts corticosteroid use and hospitalisation over 6 years of follow-up. Gut. 2016 Mar;65(3):408-14. doi: 10.1136/gutjnl-2015-309598. Epub 2015 May 18. PMID 25986946
- [Result] Rutter M, Saunders B, Wilkinson K, Rumbles S, Schofield G, Kamm M, Williams C, Price A, Talbot I, Forbes A. Severity of inflammation is a risk factor for colorectal neoplasia in ulcerative colitis. Gastroenterology. 2004 Feb;126(2):451-9. doi: 10.1053/j.gastro.2003.11.010. PMID 14762782
- [Result] Gupta RB, Harpaz N, Itzkowitz S, Hossain S, Matula S, Kornbluth A, Bodian C, Ullman T. Histologic inflammation is a risk factor for progression to colorectal neoplasia in ulcerative colitis: a cohort study. Gastroenterology. 2007 Oct;133(4):1099-105; quiz 1340-1. doi: 10.1053/j.gastro.2007.08.001. Epub 2007 Aug 2. PMID 17919486
- [Result] Korelitz BI, Sultan K, Kothari M, Arapos L, Schneider J, Panagopoulos G. Histological healing favors lower risk of colon carcinoma in extensive ulcerative colitis. World J Gastroenterol. 2014 May 7;20(17):4980-6. doi: 10.3748/wjg.v20.i17.4980. PMID 24803809
- [Result] Wiernicka A, Szymanska S, Cielecka-Kuszyk J, Dadalski M, Kierkus J. Histological healing after infliximab induction therapy in children with ulcerative colitis. World J Gastroenterol. 2015 Oct 7;21(37):10654-61. doi: 10.3748/wjg.v21.i37.10654. PMID 26457025
- [Result] Magro F, Lopes SI, Lopes J, Portela F, Cotter J, Lopes S, Moreira MJ, Lago P, Peixe P, Albuquerque A, Rodrigues S, Silva MR, Monteiro P, Lopes C, Monteiro L, Macedo G, Veloso L, Camila C, Afonso J, Geboes K, Carneiro F; Portuguese IBD group [GEDII]. Histological Outcomes and Predictive Value of Faecal Markers in Moderately to Severely Active Ulcerative Colitis Patients Receiving Infliximab. J Crohns Colitis. 2016 Dec;10(12):1407-1416. doi: 10.1093/ecco-jcc/jjw112. Epub 2016 May 25. PMID 27226417
- [Result] Fernandez-Blanco JI, Fernandez-Diaz G, Cara C, Vera MI, Olivares D, Taxonera C. Adalimumab for Induction of Histological Remission in Moderately to Severely Active Ulcerative Colitis. Dig Dis Sci. 2018 Mar;63(3):731-737. doi: 10.1007/s10620-018-4935-5. Epub 2018 Jan 25. PMID 29372480
- [Result] Steenholdt C, Brynskov J, Thomsen OO, Munck LK, Fallingborg J, Christensen LA, Pedersen G, Kjeldsen J, Jacobsen BA, Oxholm AS, Kjellberg J, Bendtzen K, Ainsworth MA. Individualised therapy is more cost-effective than dose intensification in patients with Crohn's disease who lose response to anti-TNF treatment: a randomised, controlled trial. Gut. 2014 Jun;63(6):919-27. doi: 10.1136/gutjnl-2013-305279. Epub 2013 Jul 22. PMID 23878167
- [Result] Velayos FS, Kahn JG, Sandborn WJ, Feagan BG. A test-based strategy is more cost effective than empiric dose escalation for patients with Crohn's disease who lose responsiveness to infliximab. Clin Gastroenterol Hepatol. 2013 Jun;11(6):654-66. doi: 10.1016/j.cgh.2012.12.035. Epub 2013 Jan 26. PMID 23357488
- [Result] Maser EA, Villela R, Silverberg MS, Greenberg GR. Association of trough serum infliximab to clinical outcome after scheduled maintenance treatment for Crohn's disease. Clin Gastroenterol Hepatol. 2006 Oct;4(10):1248-54. doi: 10.1016/j.cgh.2006.06.025. Epub 2006 Aug 22. PMID 16931170
- [Result] Seow CH, Newman A, Irwin SP, Steinhart AH, Silverberg MS, Greenberg GR. Trough serum infliximab: a predictive factor of clinical outcome for infliximab treatment in acute ulcerative colitis. Gut. 2010 Jan;59(1):49-54. doi: 10.1136/gut.2009.183095. PMID 19651627
- [Result] Paul S, Del Tedesco E, Marotte H, Rinaudo-Gaujous M, Moreau A, Phelip JM, Genin C, Peyrin-Biroulet L, Roblin X. Therapeutic drug monitoring of infliximab and mucosal healing in inflammatory bowel disease: a prospective study. Inflamm Bowel Dis. 2013 Nov;19(12):2568-76. doi: 10.1097/MIB.0b013e3182a77b41. PMID 24013361
- [Result] Vande Casteele N, Ferrante M, Van Assche G, Ballet V, Compernolle G, Van Steen K, Simoens S, Rutgeerts P, Gils A, Vermeire S. Trough concentrations of infliximab guide dosing for patients with inflammatory bowel disease. Gastroenterology. 2015 Jun;148(7):1320-9.e3. doi: 10.1053/j.gastro.2015.02.031. Epub 2015 Feb 24. PMID 25724455
- [Result] Cornillie F, Hanauer SB, Diamond RH, Wang J, Tang KL, Xu Z, Rutgeerts P, Vermeire S. Postinduction serum infliximab trough level and decrease of C-reactive protein level are associated with durable sustained response to infliximab: a retrospective analysis of the ACCENT I trial. Gut. 2014 Nov;63(11):1721-7. doi: 10.1136/gutjnl-2012-304094. Epub 2014 Jan 28. PMID 24474383
- [Result] Adedokun OJ, Sandborn WJ, Feagan BG, Rutgeerts P, Xu Z, Marano CW, Johanns J, Zhou H, Davis HM, Cornillie F, Reinisch W. Association between serum concentration of infliximab and efficacy in adult patients with ulcerative colitis. Gastroenterology. 2014 Dec;147(6):1296-1307.e5. doi: 10.1053/j.gastro.2014.08.035. Epub 2014 Aug 28. PMID 25173754
- [Result] Vande Casteele N, Khanna R, Levesque BG, Stitt L, Zou GY, Singh S, Lockton S, Hauenstein S, Ohrmund L, Greenberg GR, Rutgeerts PJ, Gils A, Sandborn WJ, Vermeire S, Feagan BG. The relationship between infliximab concentrations, antibodies to infliximab and disease activity in Crohn's disease. Gut. 2015 Oct;64(10):1539-45. doi: 10.1136/gutjnl-2014-307883. Epub 2014 Oct 21. PMID 25336114
- [Result] Papamichael K, Rakowsky S, Rivera C, Cheifetz AS, Osterman MT. Infliximab trough concentrations during maintenance therapy are associated with endoscopic and histologic healing in ulcerative colitis. Aliment Pharmacol Ther. 2018 Feb;47(4):478-484. doi: 10.1111/apt.14458. Epub 2017 Dec 6. PMID 29210094
- [Result] Sandborn WJ, Feagan BG, Marano C, Zhang H, Strauss R, Johanns J, Adedokun OJ, Guzzo C, Colombel JF, Reinisch W, Gibson PR, Collins J, Jarnerot G, Rutgeerts P; PURSUIT-Maintenance Study Group. Subcutaneous golimumab maintains clinical response in patients with moderate-to-severe ulcerative colitis. Gastroenterology. 2014 Jan;146(1):96-109.e1. doi: 10.1053/j.gastro.2013.06.010. Epub 2013 Jun 14. PMID 23770005
- [Result] Adedokun OJ, Xu Z, Marano CW, Strauss R, Zhang H, Johanns J, Zhou H, Davis HM, Reinisch W, Feagan BG, Rutgeerts P, Sandborn WJ. Pharmacokinetics and Exposure-response Relationship of Golimumab in Patients with Moderately-to-Severely Active Ulcerative Colitis: Results from Phase 2/3 PURSUIT Induction and Maintenance Studies. J Crohns Colitis. 2017 Jan;11(1):35-46. doi: 10.1093/ecco-jcc/jjw133. Epub 2016 Jul 20. PMID 27440869
- [Result] Detrez I, Dreesen E, Van Stappen T, de Vries A, Brouwers E, Van Assche G, Vermeire S, Ferrante M, Gils A. Variability in Golimumab Exposure: A 'Real-Life' Observational Study in Active Ulcerative Colitis. J Crohns Colitis. 2016 May;10(5):575-81. doi: 10.1093/ecco-jcc/jjv241. Epub 2016 Jan 6. PMID 26738756

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT03773445/Prot_000.pdf
  • Informed Consent Form (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT03773445/ICF_001.pdf